CLINICAL TRIAL: NCT01539343
Title: Phase II Pilot Study to Estimate the Adverse Events Associated With the Lock Solution When Used to Salvage Central Venous Catheter (CVC) in the Setting of a Central Line Associated Bloodstream Infection (CLABSI)
Brief Title: Antimicrobial Catheter Lock Solution for the Treatment of Central Line Associated Bloodstream Infection (CLABSI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Triax (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1019; NCI-2012-00302 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-02-17; First posted 2012-02-27 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Infection
Keywords: Infection; Catheter-related bloodstream infection; CRBSI; Antimicrobial Lock Therapy; ALT; Central Line Associated Bloodstream Infection; CLABSI; Central Venous Catheter; CVC; Quantitative blood cultures; QBC
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antimicrobial Lock Solution (Experimental): Participants receive the HEAL antimicrobial solution for 2 hours once daily for a minimum of 5 consecutive days. Participants also receive the lock therapy once weekly for two additional weeks. Principle ingredients include minocycline, calcium disodium ethylenediaminetetraacetate (CaEDTA) and ethanol.
  Interventions: Drug: Antimicrobial Solution

INTERVENTIONS:
Drug: Antimicrobial Solution — Antimicrobial solution, consisting of minocycline in combination with 30mg/ml of a chelator (EDTA) in 25% ethanol solution (HEAL solution), instilled in central venous catheter (CVC) catheter for 2 hours once daily for a minimum of 5 consecutive days. Lock therapy also received once weekly for two additional weeks.

SUMMARY:
A CVC is a sterile flexible tube that allows a drug to flow from a bottle or bag directly into a patient's bloodstream. CVCs may cause infections when bacteria gets into the catheter and enters the bloodstream. They also have a risk of becoming clogged. When this occurs, the CVC usually needs to be replaced.

The goal of this clinical research study is to learn if an antimicrobial catheter lock solution can make it possible for the CVC to stay in place while treating an infection with antibiotics. The safety of the solution will also be tested.

Your outcome will be compared to the outcome of patients who had the same type of infection but had their CVC removed.

The antimicrobial catheter lock solution is made up of 3 chemicals:

Minocycline and ethanol are designed to disinfect the CVC. Disodium ethylenediaminetetraacetate is designed to prevent the CVC from clogging.

DETAILED DESCRIPTION:
Study Drug Administration (Lock Solution):

If you are found to be eligible to take part in this study, the infection will be treated with antibiotics according to the standard of care. You will also receive the antimicrobial catheter lock solution through the CVC 2 hours per day for at least 5 days within the first week. In addition, you will receive the lock therapy for 2 additional days that could either be given on the following next 2 days or within the next 2 weeks. After locking the catheter for 2 hours, the HEAL lock will be cleared out, and the catheter will be flushed with normal saline and then locked with heparin or normal saline until the next time it needs to be used.

Study Visits:

On the first day after you receive the antimicrobial catheter lock solution, you will be checked for side effects such as pain, burning, discomfort, drowsiness, headache, facial redness, shortness of breath, and/or irregular heartbeat . After the last dose of receiving the catheter lock solution, you will be asked if you have experienced any side effects after receiving the catheter lock solution.

One (1) time each day while you are in the hospital, you will be checked for signs of infection and your vital signs (heart rate, breathing rate, blood pressure, and temperature) will be measured.

Every 2 days, blood (about 2 tablespoons) will be drawn to check for infection. This will continue until the blood draws no longer show signs of infection.

Every week, blood (about one teaspoon) will be drawn to check that your liver is function well.

Length of Study Participation:

You may receive the antimicrobial catheter lock solution for up to 7 days (over the course of 3 weeks). You will no longer be able to receive it if intolerable side effects occur or the infection does not go away after 7 days.

End of Treatment Visit:

* You will need to return to MD Anderson for your end of treatment visit within 7 days (+/- 3 days) after your last dose of study drug.
* At this visit, you will be asked about any symptoms or illnesses that you may have had since your last visit. You will be checked for signs of infection and your vital signs will be measured.
* Blood (about 2 tablespoons) will be drawn to check for infection. You will be asked about any antimicrobial drugs or therapies that you may be taking until the end of your treatment.

Follow-Up Visit:

You will have a follow-up visit about 1 month after receiving the last dose of antimicrobial catheter lock solution. At this visit, you will be checked for signs of infection and your vital signs will be measured. If the doctor thinks it is needed, blood (about 2 tablespoons) will be drawn to check for infection. You will be asked about any antimicrobial drugs that you may be taking until the end of your treatment.

This is an investigational study. The study lock solution is made up of minocycline, disodium ethylenediaminetetraacetate, and ethanol. Each of these are commercially available and FDA approved for other uses:

* Minocycline - for the treatment of cellulitis, acne, respiratory and urinary tract infections, gonococcal, chlamydial or ureaplasma urealyticum infections, cutaneous nocardiosis, and syphilis.
* Disodium ethylenediaminetetraacetate - for the treatment of lead poisoning
* Ethanol - for cleaning your hands

It is investigational to give minocycline, disodium ethylenediaminetetraacetate, and ethanol in combination as an antimicrobial lock solution.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older
2. Patients with indwelling CVC that have been in place for at least 14 days with documented CLABSI as defined by CDC [62]. In neutropenic patients (defined as an absolute neutrophil count (ANC) < 500 cells/mm3) with CLABSI, to confirm that CVC is the source of the bacteremia, we will use the definitions of catheter-related bloodstream infection (CRBSI) based on the mgmt guidelines of intravascular catheter related infections published by IDSA [10]. This includes the evidence that points to the CVC as the culprit: a) Paired quantitative blood cultures (QBC), whereby QBC are drawn through the CVC and peripheral vein and the blood cultures from the CVC reveal 3-fold greater number of colonies than the peripherally drawn QBC. b) Differential time to positivity, where blood cultures simultaneously drawn from the CVC and peripheral vein are positive for the same organism, and the catheter-drawn blood culture turns positive at least 2 hours earlier than the peripherally drawn blood culture.
3. Female patients must be non-lactating and at no risk for pregnancy for one of the following reasons: a) Postmenopausal for at least one year b) Post-hysterectomy and/or post-bilateral ovariectomy and/or other surgical sterilization c) If of childbearing potential, having a negative urine or serum human chorionic gonadotropin (hCG) pregnancy test within 5 days prior to study enrollment and be using a highly effective method of birth control throughout the course of the study. Reliable sexual abstinence throughout the course of the study is acceptable as a highly effective method of birth control for the purposes of this study.
4. Patients with short term non-tunneled catheters will be enrolled only if CVC cannot be removed or exchanged (patient refuses to have CVC removed, CVC needed and no other vascular access available, patient is thrombocytopenic (platelet count below 20,000) that will prohibit inserting a new CVC at a different site).

Exclusion Criteria:

1. Patients allergic to tetracycline antibiotics or calcium EDTA
2. Patients on disulfiram or disulfiram like drugs
3. Patients with severe sepsis, septic shock, hypotension or who are considered otherwise unstable
4. Presence of prosthetic valve
5. Presence of signs of metastatic deep-seated infection such as osteomyelitis or septic pulmonary infarcts or endocarditis (as evidenced by vegetations on an echocardiogram), or septic thrombosis
6. Patients with tunnel or catheter exit site infection or infusion port pocket abscess as manifested by purulence at the exit site or inflammation with erythema or induration of >1 cm in diameter.
7. Patients with Candida line infection
8. Patients who have been previously entered on the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Adverse Event Rate | 7 days
  Adverse events include symptoms of discomfort and pain associated with antimicrobial lock therapy (ALT) as well as mechanical complications. Evaluation of symptoms of discomfort related to the ALT including pain, feelings of discomfort, irritation, headache, facial redness or flushing, feeling of drowsiness, nausea, alcohol taste, dyspnea, arrhythmias. Participants given a 0 to 10 numeric discomfort scale. Toxicity due to persistent bacteremia monitored at 7 days.

SECONDARY OUTCOMES:
Resolution Efficacy of CLABSI | 1 month after treatment
  Clinical assessment pertaining to central line associated bloodstream infection (CLABSI) performed within one month from end of treatment with lock therapy. Following criteria represent infectious failure to respond: Persistent signs and symptoms associated with CLABSI (fever) after 72 hours of initiation of active systemic antimicrobial therapy. Persistent bacteremia. Relapse of bacteremia during follow-up. Development of related deep seated infections during follow-up. Infection related death during acute illness, relapse or development of related deep seated complications.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Marie Chaftari, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Raad I, Chaftari AM, Zakhour R, Jordan M, Al Hamal Z, Jiang Y, Yousif A, Garoge K, Mulanovich V, Viola GM, Kanj S, Pravinkumar E, Rosenblatt J, Hachem R. Successful Salvage of Central Venous Catheters in Patients with Catheter-Related or Central Line-Associated Bloodstream Infections by Using a Catheter Lock Solution Consisting of Minocycline, EDTA, and 25% Ethanol. Antimicrob Agents Chemother. 2016 May 23;60(6):3426-32. doi: 10.1128/AAC.02565-15. Print 2016 Jun. PMID 27001822
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org